CLINICAL TRIAL: NCT05845372
Title: Association of Prophylactic Use of Stress Ulcer Drugs and Clinical Outcomes in Patients With Acute Anterior Circulation Thrombectomy: a Prospective, Multicenter, Observational Cohort Study
Brief Title: Association of Prophylactic Use of Stress Ulcer Drugs and Clinical Outcomes in Patients With Acute Anterior Circulation Thrombectomy
Status: Not yet recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Guangzhou Medical University (Other); The Affiliated Hospital of Inner Mongolia Medical University (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); Second Affiliated Hospital of Guangxi Medical University (Other); Fujian Medical University Union Hospital (Other); Huizhou Municipal Central Hospital (Other); Haikou People's Hospital (Other); Kashgar 1st People's Hospital (Other); Ganzhou City People's Hospital (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Huadu District People's Hospital of Guangzhou (Other); Dongguan donghua hospital (Unknown); Sinopharm North Hospital (Unknown); Heyuan people's Hospital (Unknown); Hainan People's Hospital (Other); Hainan Traditional Chinese Medicine Hospital (Unknown); The First Affiliated Hospital of Hunan University of Traditional Chinese Medicine (Other); The Second Hospital University of South China (Other); Dongguan People's Hospital (Other Government); Yueyang People's Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: NFEC-2023-040
Record Dates: First submitted 2023-04-26; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute Ischemic Stroke; Stress Ulcer Bleeding; Mechanical Thrombectomy
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stress Ulcer Prophylaxis: Subjects are on stress ulcer medications including PPIs, H2RBs, and mucosal protectors at 24 h of admission.
- Control Group: Subjects are not on stress ulcer medications including PPIs, H2RBs, and mucosal protectors at 24 h of admission.

SUMMARY:
Ischemic stroke accounts for a relatively high proportion of strokes. In recent years, intravenous thrombolysis and endovascular therapy have significantly improved the revascularization rate in patients with large vessel occlusive cerebral infarction, but 20-50% of patients still experience ineffective revascularization. Therefore, postoperative monitoring and treatment of patients with large vessel occlusions is crucial for early recognition, management and prevention of complications. Stress ulcer bleeding is a serious complication after acute ischemic stroke, with a prevalence of 1%-5%, and a previously proven incidence of stress ulcer bleeding after ischemic stroke. Stress ulcer bleeding after ischemic stroke has been shown to be closely associated with unfavorable outcomes, such as mortality. Current national and international guidelines or consensus on the prevention of stress ulcers after acute ischemic stroke do not advocate the routine use of histamine receptor antagonists or proton pump inhibitors for the prevention of stress ulcers, but rather should be considered in the context of the patient's risk factors for stress ulcers and discontinued after the patient initiates enteral nutrition. However, there is no evidence-based medical evidence to support the risk-benefit relationship of stress ulcer drug prophylaxis in patients with mechanical thrombectomy for acute anterior circulation large vessel occlusion.

DETAILED DESCRIPTION:
Stress ulcer bleeding is a serious complication after acute ischemic stroke, with a prevalence of 1%-5%, of which only 0.5%-1% require blood transfusion or result in hypotension. Stress ulcer bleeding after ischemic stroke has been shown to be associated with poor outcomes, such as mortality, and basilar artery occlusion and middle cerebral artery cerebral infarction are independent risk factors for stress ulcer bleeding after acute ischemic stroke. Guidelines or consensus on the prevention of stress ulcers after acute ischemic stroke do not advocate the routine use of histamine receptor antagonists or proton pump inhibitors for stress ulcer prevention.

However, stress ulcer prophylaxis is initiated in most patients admitted to the neurological intensive care unit after mechanical embolization of acute anterior circulation large vessel occlusion. With advances such as diagnosis and early initiation of enteral nutrition, the rate of stress ulcer bleeding in patients with mechanical embolization of acute anterior circulation large vessel occlusion is significantly reduced. The relationship between the risk and benefit of SUP in patients undergoing mechanical embolization for acute anterior circulation large vessel occlusion is not yet supported by evidence-based medical evidence. Therefore, the purpose of this study was to investigate the correlation between pharmacological stress ulcer prophylaxis and clinical outcomes in patients undergoing mechanical thrombectomy for acute anterior circulation large vessel occlusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Within 24 hours of onset. Meet the criteria for diagnosis of acute ischemic stroke in the "China Acute Ischemic Stroke Diagnosis and Treatment Guidelines 2018".
3. Meet the indications for mechanical thrombectomy in the "Chinese Guidelines for Early Endovascular Interventions in Acute Ischemic Stroke 2022".
4. Treated with mechanical thrombectomy.
5. NIHSS score ≥ 6 at onset of illness.
6. Sign an informed notice.

Exclusion Criteria:

Allergy to drug ingredients. Women who are pregnant or breastfeeding. Life expectancy of less than 3 months due to other non-ischemic stroke diseases such as malignancy, severe liver or renal failure.

Have participated in other interventional clinical studies (affecting the outcome of this cohort study).

Participants who were judged by the investigator to be unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are treated with mechanical thrombectomy with acute anterior circulation large vessel occlusion. ≥18 years of age, within 24 hours of onset. Expected survival >3 months. NIHSS score ≥ 6 at onset of illness.
Sampling Method: Probability Sample
Enrollment: 2592 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
90-day mortality after onset | 90-day after onset
  Proportion of enrolled patients who died 90 days after onset of disease.
Incidence of stroke-associated pneumonia | within 7-day of onset
  Incidence of non-mechanically ventilated stroke patients with new pneumonia within 7-day of onset

SECONDARY OUTCOMES:
Incidence of clinically significant bleeding | within 7-day of onset
  One of the following 4 symptoms occurs within 24 hours of bleeding from a stress ulcer (in the absence of other causes):1. A decrease of ≥ 20 mmHg in any one of systolic, diastolic and mean arterial pressure. 2.Initiation of blood pressure boosters or 20% increase in medication dose.3. Decreased hemoglobin ≥ 2 g/d(（1.24 mmol/l). 4.Infusion of erythrocytes ≥ 2 U.
Incidence of stress ulcer bleeding | 7-day after onset
  Coffee-like residue/black stool/blood in stool within 7-day after onset and more than 2 consecutive positive fecal/gastric fluid occult blood
Incidence of unfavorable functional prognosis at 90 days after onset | 90-day after onset
  Incidence of unfavorable functional prognosis at 90 days after onset
90-day mRS score change | 90-day after onset
  Modified Rankin Scale score change within 90 days after onset in patients who were eligible for inclusion criteria
Incidence of early neurological deterioration | within 72 hours after onset
  Increased score of National Institutes of Health Stroke Scale within 72h after onset ≥ 4
1-year post-onset mortality | 1 year after onset
  Mortality at 1 year after onset in patients who were eligible for inclusion criteria
Incidence of adverse related events such as pneumonia or myocardial ischemia 1 year after onset | 1 year after onset
  Incidence of adverse related events such as pneumonia or myocardial ischemia 1 year after onset in patients who were eligible for inclusion criteria

CONTACTS AND LOCATIONS:
Overall Officials: Suyue Pan, Principal Investigator — Department of Neurology, Nanfang Hospital,Southern Medical University
Locations (19):
- China (19):
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Dongguan donghua hospital, Dongguan, Guangdong
  - Dongguan People's Hospital, Dongguan, Guangdong
  - Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong
  - Huadu District People's Hospital of Guangzhou, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Fourth Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Heyuan people's Hospital, Heyuan, Guangdong
  - Huizhou Municipal Central Hospital, Huizhou, Guangdong
  - Haikou People's Hospital, Haikou, Hainan
  - Hainan Provincial People's Hospital, Haikou, Hainan
  - Hainan Traditional Chinese Medicine Hospital, Haikou, Hainan
  - The First Hospital of Changsha, Changsha, Hunan
  - The Second Hospital University of South China, Hengyang, Hunan
  - Yueyang People's Hospital, Yueyang, Hunan
  - Sinopharm North Hospital, Baotou, Inner Mongolia
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Ganzhou City People's Hospital, Ganzhou, Jiangxi
  - Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang